CLINICAL TRIAL: NCT06915831
Title: Obstructive Sleep Apnea and Glycemic Dysregulation in Adults With Type 1 Diabetes
Brief Title: Type 1 Diabetes and Obstructive Sleep Apnea
Acronym: T1D and OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB24-2170; 1R01HL174685-01 (NIH)
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Sleep Apnea, Obstructive; Type 1 Diabetes (T1D)
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus, Type 1 | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Within subjects design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Untreated (No Intervention): No treatment for OSA
- Treated: Continuous positive airway pressure (CPAP) treatment (Active Comparator): Treatment for OSA by CPAP
  Interventions: Device: Continuous positive airway pressure (CPAP)

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) — All-night CPAP will be applied with bedtimes 23:00h to 7:00h.
  Arms: Treated: Continuous positive airway pressure (CPAP) treatment

SUMMARY:
The purpose of the study is to investigate the role of sleep apnea in glycemic dysregulation in adults with Type 1 diabetes.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common sleep disorder characterized by recurrent collapse of upper airway during sleep, resulting in intermittent hypoxia, sleep fragmentation by transient arousals, and poor sleep quality. Continuous positive airway pressure (CPAP), applied at night, is considered the treatment of choice for persons who are diagnosed with OSA. Current evidence suggests that OSA is highly prevalent in adults with T1D and particularly those with moderate-to-severe OSA have poorer glycemic control. Our overall goal is to investigate the role OSA in glycemic dysregulation in adults with T1D.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 50 years old
* Type 1 Diabetes on insulin pump therapy and using a CGM device with an GMI (glucose management indicator) between 5.5 and 8.5% with hemoglobin in the normal range at screening
* OSA by home sleep apnea test

Exclusion Criteria:

* Regular and adherent CPAP use per clinical guidelines
* Requiring oxygen or advanced positive airway pressure modalities during sleep
* Having a 'fall-asleep' or 'near miss' accident in the past 6-months
* Shift work
* Severe hypoglycemia (≥1 episode in the past 3 months or diagnosis of hypoglycemic unawareness)
* ≥1 trip to emergency room for poor glucose management in the past 6 months
* Proliferative retinopathy
* Fasting triglycerides >400mg/dL,
* Liver transaminases >2 times upper limit of normal,
* Renal transplantation or serum creatinine >1.5 mg/dL
* Anemia (hemoglobin <13.0g/dL in men or <11.6g/dL in women)
* Acute coronary syndrome or stroke past 6 months
* Severe hypertension (blood pressure>180/105 mmHg)
* Any other significant health condition: unstable angina, heart failure requiring hospitalization in the past 6 months, significant heart block or arrhythmias, NYHA Class>2, pulmonary disease with dependence on oxygen or daily use of bronchodilators, active or chronic infection, thyroid disease and other endocrine disorders (e.g. Cushing syndrome, acromegaly)
* Recent major surgery
* Major psychiatric disorder
* Subjects will also be excluded if taking medications that can confound metabolic assessments including systemic glucocorticoids, antipsychotics, thiazide diuretics, beta-blockers, daily use of aminophylline or theophylline, or use of any immunosuppressant.
* Currently pregnant or trying to get pregnant or nursing
* Smoking, alcohol or illegal drug abuse

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic variability | Within 3 months of screening
  Glycemic variability will be calculated using a standard metric as percent coefficient of variation (% CV) of glucose values obtained from continuous glucose monitoring (CGM).

CONTACTS AND LOCATIONS:
Overall Officials: Esra Tasali, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT06915831/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT06915831/ICF_001.pdf